CLINICAL TRIAL: NCT00370032
Title: A Randomize, Placebo-controlled, Crossover Study to Measure the Effect of Alosetron on Mucosal Blood Flow in Female Healthy Volunteers and Diarrhea-predominant IBS Subjects
Brief Title: Study to Assess the Effect Of Alosetron On Mucosal Blood Flow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: S3B40042
Record Dates: First submitted 2006-08-28; First posted 2006-08-30 (Estimated); Results first posted 2009-04-02 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Irritable Colon
Keywords: mucosal blood flow d-IBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — alosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: alosetron

SUMMARY:
This study will look at colonic mucosal blood flow in subjects who have taken alosetron vs placebo and healthy volunteers vs diarrhea-predominant Irritable Bowel Syndrome (d-IBS) patients.

ELIGIBILITY:
Inclusion criteria:

* The subject signs and dates a written informed consent form prior to the initiation of any study-related activities.
* The subject is between 18 and 49 years of age at the time of the Screening Visit.
* The subject is female and either:

  * A healthy subject. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history (including family), physical examination, laboratory studies, and other tests.

OR

* A d-IBS patient per the Rome II criteria who has a normal result from a flexible sigmoidoscopy or colonoscopy, or flexible sigmoidoscopy plus barium enema, within 2 years of the Screening visit.

  * The subject demonstrates a negative urine pregnancy test result prior to investigational product administration and be either:
* Of non-childbearing potential (i.e., physiologically incapable of becoming pregnant)
* post-menopausal define as one year without menses in the absence of hormone replacement therapy.
* sterilization (via hysterectomy or bilateral tubal ligation)
* Of childbearing potential and agrees to one of the following acceptable non-hormonal contraceptive methods consistently and in accordance with both the product label and the instructions of a physician. Subjects will use effective contraceptive methods for at least one month prior to Screening and should continue to use the same contraceptive method throughout the study (Follow-up Visit).
* Complete abstinence from intercourse
* an intra-uterine device (IUD) inserted by a qualified physician, provided the IUD is not of the hormonal type and it has published data showing that the highest expected failure rate is less than 1% per year (not all IUDs meet this criterion)
* double barrier method if comprised of a spermicide with either a condom or diaphragm
* sterilization of partner The subject is ambulatory (defined as not depending exclusively on a wheelchair for mobility).

Exclusion criteria:

* The subject is taking oral contraceptive or other hormonal therapy.
* The subject has a concurrent illness or disability that may affect the interpretation of clinical data, or otherwise contraindicates participation in this clinical study (e.g., an unstable cardiovascular, autoimmune, renal, hepatic, pulmonary, endocrine, metabolic, gastrointestinal, hematologic, or neurological condition).
* The subject has constipation-predominant IBS (c-IBS) or alternating IBS per the ROME II criteria.
* The subject has current evidence of or history of chronic or severe constipation, or a history of sequelae from constipation.
* Evidence of a biochemical or structural abnormality of the digestive tract. These conditions include (but not limited to):

  * Current evidence, or history of (at any time in the past):
  * GI/Bowel conditions:
  * inflammatory bowel disease (Crohn's disease or ulcerative colitis)
  * celiac disease
  * laxative abuse (in the clinical judgement of the physician)
  * gastrointestinal surgery (exceptions include ≥6 months post-surgery appendectomy, cholecystectomy, fundoplication without gas bloat, or hiatal hernia repair; ≥3 months post-surgery herniorrhaphy without bowel resection)
  * gastroparesis
  * GI malignancy
  * carcinoid syndrome
  * amyloidosis
  * gastrointestinal adhesions
  * ischemic colitis
  * toxic megacolon
  * impaired intestinal circulation
  * gastrointestinal perforation
  * gastrointestinal obstruction and/or stricture
  * Ischemic cardiovascular conditions:
  * coronary artery disease (CAD)
  * significant atherosclerosis
  * chronic pancreatitis
  * diabetes
  * thrombophlebitis or hypercoagulable state.
  * Current evidence of (within the past 6 months):
  * diverticulitis
  * ileus
  * symptomatic cholelithiasis
  * proctitis.
  * Current evidence of:
  * Hemoccult (+) stool.
* The subject has a BMI of ≥27.
* Mental impairment or inability or refusal to follow directions.
* The subject has current evidence of, or has been treated for a malignancy within the past five years (other than localized basal cell, squamous cell skin cancer or cancer in situ that has been resected).
* The subject exhibits evidence of hepatic dysfunction, viral hepatitis, or exhibits serum ALT (alanine aminotransferase) (SGPT), AST (aspartate aminotransferase) (SGOT) values >2.5 times the upper limit of normal or alkaline phosphatase or bilirubin values >2.0 times the upper limit of normal.
* The subject displays renal impairment as evidenced by a serum creatinine value >2.0 mg/dl.
* The subject has used any medication within the seven days prior to dosing, unless approved by the investigator and GlaxoSmithKline (GSK) personnel. Section 9.1.
* The subject has used an investigational drug, or participated in an investigational study, within 30 days of the Screening Visit.
* The subject has a history of drug allergies (including but not limited to hypersensitivity responses to alosetron which, in the opinion of the investigator, contraindicates the subject's participation in this study.
* Subjects who have made a blood donation (>450mL) within 6 weeks prior to screening.
* The subject has a history of alcohol and/or substance abuse within the past two years.
* The subject is pregnant. The subject is breastfeeding.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- d-IBS (Diarrhea Predominant - Irritable Bowel Syndrome): Subjects with diarrhea-predominant irritable bowel syndrome. This group was randomize to EITHER 0.5 mg BID Alosetron or Placebo for 6 days followed by a flexible sigmoidoscopy; followed by a 7 day washout period; Then the subjects who were given study drug the first treatment period were given Placebo and vice versa for the next 6 days followed by a flexible sigmoidoscopy then had a 7 day follow up period.
- Healthy Volunteers: Subjects with no clinical disease. This group was randomize to EITHER 0.5 mg BID Alosetron or Placebo for 6 days followed by flexible sigmoidoscopy then had a 7 day washout period; Then the subjects who were given study drug the first treatment period were given Placebo and vice versa for the next 6 days followed by another 7 day wash out period and a 7 day follow up period.
Period: Treatment Period 1
Arm/Group | d-IBS (Diarrhea Predominant - Irritable Bowel Syndrome) | Healthy Volunteers
Started | 24 (Safety Population - all subjects who took at least one dose of study medication.) | 25 (Safety Population - all subjects who took at least one dose of study medication.)
Completed | 24 | 24
Not Completed | 0 | 1
Not completed — Unable to perform sigmoidoscopy on Day 6 | 0 | 1
Period: Washout Period
Arm/Group | d-IBS (Diarrhea Predominant - Irritable Bowel Syndrome) | Healthy Volunteers
Started | 24 | 24
Completed | 23 | 22
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 0
Period: Treatment Period 2
Arm/Group | d-IBS (Diarrhea Predominant - Irritable Bowel Syndrome) | Healthy Volunteers
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0
Period: Follow-up Period
Arm/Group | d-IBS (Diarrhea Predominant - Irritable Bowel Syndrome) | Healthy Volunteers
Started | 23 | 22
Completed | 22 | 22
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- d-IBS: Diarrhea-predominant irritable bowel syndrome. This group was randomize to EITHER 0.5 mb BID Alosetron or Placebo for 6 days followed by a flexible sigmoidoscopy; followed by a 7 day washout period; Then the subjects who were given study drug the first treatment period were given Placebo and vice versa for the next 6 days followed by another wash out period and a 7 day follow up period.
- Healthy Volunteers: Volunteers without clinical disease. This group was randomize to EITHER 0.5 mb BID Alosetron or Placebo for 6 days followed by a flexible sigmoidoscopy; followed by a 7 day washout period; Then the subjects who were given study drug the first treatment period were given Placebo and vice versa for the next 6 days followed by another wash out period and a 7 day follow up period.
- Total: Total of all reporting groups
Arm/Group | d-IBS | Healthy Volunteers | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (8.8) | 26.9 (5.8) | 29.99 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian/European | 17 | 16 | 33
  African American | 3 | 2 | 5
  Central/South Asian | 1 | 1 | 2
  East Asian | 1 | 0 | 1
  South East Asian | 0 | 2 | 2
  Mixed Race | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Left Colon Mucosal Blood Flow (MBF)
Description: On Day 6 of each treatment period; 1 hour after dosing, subjects underwent a flexible sigmoidoscopy with Laser Doppler Flowmetry (LDF) to measure Mucosal Blood Flow (MBF). There were no pre-treatment LDF procedure, MBF was compared between the Healthy volunteers and D-irritable bowel syndrome (IBS) cohorts using the flow rates from the placebo treatment period.
Time Frame: Day 6 after each treatment period
Population: Per Protocol Population - the population used for the primary and secondary outcome analyses. The population consisted of all randomized subjects who completed the study with MBF measurements for both treatment periods.
Measure: Mean (Standard Deviation); unit: ml per minute per 100 grams of tissue
Groups:
- d-IBS Placebo: Subjects with diarrhea-predominant irritable bowel syndrome. In Treatment Period 1 this group was first randomized to Placebo for 6 days followed by a flexible sigmoidoscopy; followed by a 7 day washout period; Then, in Treatment Period 2 the subjects were given Alosetron 0.5 mg (BID)for 5 days and on the 6th day one dose and a flexible sigmoidoscopy; followed by another wash out period of 7 days and a 7 day follow up period.
- d-IBS Alosetron: Subjects with diarrhea-predominant irritable bowel syndrome. In Treatment Period 1, this group was randomized to 0.5 mb BID Alosetron for 5days and 1 dose on the 6th day followed by a flexible sigmoidoscopy; followed by a 7 day washout period; Then, in Treatment Period 2 the subjects were given Placebo for the next 6 days followed by another 7 day wash out period and a 7 day follow up period.
- Healthy Volunteers Placebo: Subjects without Clinical disease. In Treatment Period 1 this group was first randomized to Placebo for 6 days followed by a flexible sigmoidoscopy; followed by a 7 day washout period; Then, in Treatment Period 2 the subjects were given Alosetron 0.5 mg (BID)for 5 days and on the 6th day one dose and a flexible sigmoidoscopy; followed by another wash out period of 7 days and a 7 day follow up period.
- Healthy Volunteers Alosetron: Subjects without clinical disease. In Treatment Period 1 this group was randomized to 0.5 mb BID Alosetron for 5days and 1 dose on the 6th day followed by a flexible sigmoidoscopy; followed by a 7 day washout period; Then,in Treatment Period 2 the subjects were given Placebo for the next 6 days followed by another 7 day wash out period and a 7 day follow up period.
Arm/Group | d-IBS Placebo | d-IBS Alosetron | Healthy Volunteers Placebo | Healthy Volunteers Alosetron
Number analyzed (Participants) | 22 | 22 | 19 | 19
ml per minute per 100 grams of tissue | 125.6 (38.6) | 117.5 (37.71) | 130.7 (40.12) | 121.6 (51.26)
Statistical Analysis 1: Comparison: d-IBS Placebo vs d-IBS Alosetron; Test type: Superiority or Other; p = 0.131, paired t-test Hommel-Simes; Mean Difference (Final Values) = -8.1, 95% CI [-18.4 to 2.157]
Statistical Analysis 2: Comparison: Healthy Volunteers Placebo vs Healthy Volunteers Alosetron; Test type: Superiority or Other; p = 0.131, paired t-test Hommel-Simes; Mean Difference (Final Values) = -9.11, 95% CI [-21.2 to 2.997]

2. Secondary Outcome: Rectal Mucosal Blood Flow (MBF)
Description: On Day 6 of each treatment period approximately 1 hour after dosing, subjects underwent a flexible sigmoidoscopy with Laser Doppler Flowmetry (LDF) to measure Mucosal Blood Flow (MBF). There was no pre-treatment LDF procedure, MBF was compared between the Healthy and d-IBS cohorts using the flow rates from the placebo treatment period.
Time Frame: Day 6 after each treatment period
Measure: Mean (Standard Deviation); unit: ml per minute per 100 grams of tissue
Groups:
- d-IBS Alosetron: Subjects with diarrhea-predominant irritable bowel syndrome. In Treatment Period 1 this group was randomized to 0.5 mb BID Alosetron for 5days and 1 dose on the 6th day followed by a flexible sigmoidoscopy; followed by a 7 day washout period; Then, in Treatment Period 2 the subjects were given Placebo for the next 6 days followed by another 7 day wash out period and a 7 day follow up period.
Arm/Group | d-IBS Placebo | d-IBS Alosetron | Healthy Volunteers Placebo | Healthy Volunteers Alosetron
Number analyzed (Participants) | 22 | 22 | 22 | 22
ml per minute per 100 grams of tissue | 173 (45.52) | 159.1 (51.73) | 149.1 (39.82) | 140.3 (56)

3. Secondary Outcome: Left Colon and Rectal Mucosal Blood Flow Cohort Comparisons
Description: as for outcome 2
Time Frame: Day 6 after each treatment period
Population: Population: modified per protocol to include placebo information only.
Measure: Mean (Standard Deviation); unit: ml per minute per 100 grams of tissue
Groups:
- d-IBS Placebo - Left Colon: Subjects with diarrhea-predominant irritable bowel syndrome . Modified per protocol. Subjects Left Colon Mucosal blow flow under placebo.
- d-IBS Placebo - Rectal: Subjects with diarrhea-predominant irritable bowel syndrome. Modified per protocol. Subjects Rectal Mucosal blow flow under placebo.
- Healthy Volunteers Placebo - Left Colon: Subjects without Clinical disease. Modified per protocol. Subjects Left Colon Mucosal blow flow under placebo.
- Healthy Volunteers Placebo - Rectal: Subjects without clinical disease. Modified per protocol. Subjects Rectal Mucosal blow flow under placebo.
Arm/Group | d-IBS Placebo - Left Colon | d-IBS Placebo - Rectal | Healthy Volunteers Placebo - Left Colon | Healthy Volunteers Placebo - Rectal
Number analyzed (Participants) | 22 | 22 | 19 | 22
ml per minute per 100 grams of tissue | 135.1 (38.6) | 178.9 (45.52) | 149.9 (40.12) | 166.6 (39.82)

ADVERSE EVENTS:
Groups:
- d-IBS Placebo: Diarrhea-predominant irritable bowel syndrome. Participants receiving 0.5 mb Placebo BID in either the first or second 6-day treatment period. Both treatment periods were followed by a 7-day washout period; the second washout period was followed by a 7-day follow up period.
- d-IBS Alosetron: Diarrhea-predominant irritable bowel syndrome. Participants receiving 0.5 mb Alosetron BID in either the first or second 6-day treatment period. Both treatment periods were followed by a 7-day washout period; the second washout period was followed by a 7-day follow up period.
- Healthy Volunteers Placebo: Volunteers without clinical disease. Participants receiving 0.5 mb Placebo BID in either the first or second 6-day treatment period. Both treatment periods were followed by a 7-day washout period; the second washout period was followed by a 7-day follow up period.
- Healthy Volunteers Alosetron: Volunteers without clinical disease. Participants receiving 0.5 mb Alosetron BID in either the first or second 6-day treatment period. Both treatment periods were followed by a 7-day washout period; the second washout period was followed by a 7-day follow up period.
Arm/Group | d-IBS Placebo | d-IBS Alosetron | Healthy Volunteers Placebo | Healthy Volunteers Alosetron
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 12/24 | 10/23 | 11/24 | 11/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | d-IBS Placebo (N=24) | d-IBS Alosetron (N=23) | Healthy Volunteers Placebo (N=24) | Healthy Volunteers Alosetron (N=23)
Abdominal Distention (Gastrointestinal disorders) | 1 | 0 | 1 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 4 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 3 | 3 | 2
Acarodermatitis (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 3 | 3
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.